CLINICAL TRIAL: NCT07021586
Title: Tongue Pressure in Middle-Aged and Elderly Individuals With Chronic Cervical Pain
Status: Recruiting | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yi-Fen Shih, Professor, Department of Physical Therapy and Assistive Technology, National Yang Ming Chaio Tung University, National Yang Ming Chiao Tung University
Other Study IDs: NYCU113186AE
Record Dates: First submitted 2025-05-21; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-11

CONDITIONS: Cervical Pain, Posterior; Swallowing Difficulties; Swallowing Disorders
MeSH Terms: conditions — Neck Pain; Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
The goal of the cross-sectional study is to explore the impact of neck pain on tongue pressure in the middle-aged and elderly population and analyze the effects of different cranio-cervical positioning on tongue pressure performance.

The main questions it aims to answer are:

1. Do middle-aged and elderly individuals with chronic cervical pain exhibit reduced maximal tongue pressure compared to those without cervical pain?
2. What are the effects of different cranio-cervical positioning on tongue pressure performance?

Participants will complete all the assessments on the day of testing.

DETAILED DESCRIPTION:
1. For Quality assurance plan that addresses data validation and registry procedures:

(1) Relevant data will be recorded by the researchers. All assessments will be conducted in the Orthopedic Laboratory at National Yang Ming Chiao Tung University, where the equipment is regularly maintained and monitored.

2. For Standard operating procedures to address registry operations and analysis activities:

(1 ) Participants will be recruited from clinics and communities in the Taipei and New Taipei City. Collected data will include personal information such as height, age, weight, and the number of removable dentures. Data management and analysis will be conducted using laboratory-designated computers for data storage and processing. Any adverse events, such as throat or tongue soreness occurring within 1-2 days after testing, will be recorded and reported to the researchers.

3. For Sample size assessment:

(1) Total forty participants aged between 50-65 years.

4. For missing data:

(1) This study is a cross-sectional, single-session assessment, and therefore the likelihood of missing data is minimal and no specific handling procedures are needed.

5. For statistical analysis:

(1) Data analysis for this study was conducted using SPSS software version 29.0. Continuous and categorical variables were compared between the two groups using independent t-tests and chi-square tests. Other outcomes will be analyzed using two-way mixed ANOVA, independent t-tests, or Pearson's correlation coefficient to compare differences between groups or examine associations. The significance level is set at 0.05, with p-values less than 0.05 considered statistically significant.

ELIGIBILITY:
1. Inclusion Criteria (chronic cervical pain group):

1. Aged between 50-65 year olds
2. Chronic neck pain (caused by specific neck movements or prolonged neck posture)
3. Cervical pain duration: at least 3 months within the past year
4. Cervical pain intensity: during activity or rest, as measured by the Numeric Pain Rating Scale, must have an average score of at least 3 over the past two weeks
5. No anti-inflammatory or painkillers can be used within 48 hours prior to the test

2. Inclusion Criteria (healthy group):

1. Matching gender, age, and body mass index with those in the chronic cervical pain group
2. No cervical pain has occurred within the past 6 months

3. Exclusion Criteria:

1. Neurological diseases that may affect tongue pressure readings, such as stroke or Parkinson's disease
2. Head or neck surgery in the past year
3. Severe head or neck injuries (e.g., whiplash from a car accident) in the past year
4. Diagnosed with cervical radiculopathy or myelopathy with symptoms in the form of numbness or tingling, or fail relative clinical tests (spurling's/ cervical distraction/ cervical rotation test/ upper limb tension test-1/ Hoffman sign)
5. History of head or neck deformities or cancer
6. History of head or neck radiation therapy
7. Diagnosed with dysphagia
8. Experience pain or restricted movement in the temporomandibular joint (TMJ) during chewing in the last 6 months
9. Require anticonvulsants or antidepressant medications
10. Cognitive impairments preventing understanding of the test order or communication

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community and regional clinics in Taipei or New Taipei
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximal tongue pressure | Because it is a cross sectional study with one-time measurement, it usually take five minutes to collect the data.
  Tongue pressure is used to measure the function or strength of the tongue. The higher the value, the greater the tongue strength. The measurement unit is kPa, with 0 being the minimum value. It tends to decrease with age, typically with 60 years old as the cutoff. For those under 60, the value is around 40 kPa, and for those over 60kPa, it decreases to around 33 kPa. Additionally, when accompanied by other conditions, such as dysphagia or sarcopenia, the decline is more pronounced.

SECONDARY OUTCOMES:
Mandarin version of Eating Assessment Tool-10 | It usually take 5-10 minutes to finish the questionnaire
  The Eating Assessment Tool is a commonly used self-administered questionnaire for screening potential swallowing difficulties. In this study, the Mandarin version of the EAT-10 is utilized. The questionnaire consists of 10 items, where participants rate the severity of their swallowing-related symptoms based on their subjective perception. Each item is scored from 0 (no problem) to 4 (severe problem), with a total possible score of 40. Higher scores indicate greater severity of perceived swallowing difficulties.
Repetitive Saliva Swallowing Test | It usually take 30 seconds to collect the data.
  Repetitive Saliva Swallowing Test is a simple and relatively safe test used to screen for potential functional swallowing difficulties. During the test, the participant first moistens their mouth with water. The examiner places their index finger under the participant's tongue and their middle finger on the participant's laryngeal prominence. The test instruction is, 'Please swallow saliva as much as possible until I say stop.' The examiner palpates the participant's laryngeal prominence to feel the movements during swallowing and counts the number of swallows. The test duration is 30 seconds. If the participant swallows less than three times within 30 seconds, it is used as the screening criterion for potential functional swallowing difficulty.
Temporomandibular joint kinematics | Because it is a cross sectional study with one-time measurement, it usually take twenty minutes to collect the data.
  Temporomandibular joint kinematics is used to measure the kinematics of the temporomandibular joint. The parameters include maximal mouth opening, left/right mandibular deviation, protrusion, left/right total condylar length path, and left/right total condylar translation, with measurements in millimeters (mm). Left/right total condylar rotation is measured in degrees. A larger value for the above parameters indicates greater temporomandibular joint mobility.
Craniovertebral angle | Because it is a cross sectional study with one-time measurement, it usually take five minutes to collect the data.
  The craniovertebral angle is defined as the acute angle formed by the intersection between two lines: one is the horizontal line passing through the spinous process of the seventh cervical vertebra, and the other is the line connecting the seventh cervical vertebra and the tragus of the ear. If this angle is less than 50 degrees, it is defined as exhibiting a forward head posture. The smaller the angle, the more severe the forward head posture.
Maximal handgrip strength | It usually take five minutes to collect the data.
  This study uses a digital hand dynamometer to measure maximal grip strength. A higher value indicates greater handgrip strength. When the handgrip strength is less than 28 kg for males or less than 18 kg for females, it suggests a potential tendency for sarcopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Fen Shih, Study Chair — National Yang Ming Chiao Tung University
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan